CLINICAL TRIAL: NCT05315765
Title: Development of a Patient Reported Outcome Measure for GastroIntestinal Recovery
Acronym: PRO-diGI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH20670; NIHR 201492 (Other Grant/Funding Number: National Institute for Health Research RfPB)
Record Dates: First submitted 2021-10-07; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Ileus; Small Bowel Obstruction; Intestinal Failure
Keywords: PROM; surgery
MeSH Terms: conditions — Ileus; Intestinal Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phase 1: Qualitative interviews with patients to generate thematic framework and questionnaire
- Phase 2: Face validity assessment of questionnaire
- Phase 3: Completion of questionnaire to refine scale and item list

SUMMARY:
People who undergo surgery, or develop intestinal obstruction will spend a period of time without normal bowel function. This might extend beyond the normal measures of passage of flatus or tolerance of diet. This study will take a three stage approach to develop a patient reported outcome measure for gastrointestinal recovery.

Stage 1: Qualitative interviews with 20-40 patients who have undergone major abdominal surgery, or conservatively managed intestinal obstruction. These interviews will identify key themes and ideas to develop the questionnaire.

Stage 2: Face validity testing of questionnaire with 20 patients, using the QQ-10 questionnaire to aid assessment. The questionnaire may be edited after this.

Stage 3: 250-500 patients will be asked to complete the questionnaire following surgery or treatment for intestinal obstruction. Basic demographics will also be collated. Item reduction and scale refinement will be undertaken using this dataset. This will provide a PROM of gastrointestinal recovery which is ready for validation.

DETAILED DESCRIPTION:
Gastrointestinal dysfunction is commonly seen after surgery, and also manifests itself in intestinal obstruction. During this time, the patient may experience a range of symptoms of acute intestinal failure, including loss of motility and absorption. These may resolve at different rates during the period of gastrointestinal recovery. Trials in the area have conflicting results, partly due to the selection of clinician reported unidimensional outcomes. There is a clear need for a patient reported outcome measure (PROM) to record gastrointestinal recovery.

Aims and Objectives

* To develop a PROM for gastrointestinal recovery.
* To identify a candidate long-list of items for inclusion in a PROM through semi-structured patient interviews, and test face validity with patients and an expert panel
* To develop a PROM using the approved long list

Methods This study will be conducted in three stages with reference to FDA (Food and Drug Administration) and ISOQoL (International Society for Quality of Life Research) guidelines.

Stage 1: Five centres will undertake purposive sampling to identify patients who have undergone major intraabdominal surgery (including gastrointestinal, urological, and gynaecological) and patients treated for intestinal obstruction. It is expected that 40-60 participants will undergo a semi-structured interview to identify important items related to recovery of gastrointestinal function in order to reach thematic saturation. Interviews will be transcribed and coded using a framework methodology. This will generate allow us to construct a prototype questionnaire with an initial pool of items.

Stage 2: The prototype questionnaire will be shown to a group of international experts in gastrointestinal recovery for assessment of face validity, using the QQ-10 (Questionnaire quality-10 item) questionnaire. This will then be tested with 20 patients treated for eligible conditions at five participating centres using the QQ-10.

Stage 3: Upto 500 participants (depending on number of items on the questionnaire) will be recruited from 10 centres which offer gastrointestinal, urological, and gynaecological surgery. Participants will rate items on a Likert scale. Items will undergo factor analysis to reduce the number of items. This will present a shorter questionnaire with finalised scales.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (aged 18+) admitted to hospital for one of the following reasons will be eligible to participate:

* Undergoing major elective gastrointestinal surgery (e.g. colorectal resection, gastric resection, liver or pancreatic resection)
* Emergency laparotomy for non-trauma indication
* Patients undergoing intra-abdominal surgery for non-gastrointestinal indications e.g.cystoprostatectomy, prostatectomy, nephrectomy, hysterectomy, or oophorectomy.
* With a diagnosis of intestinal obstruction (small or large bowel).
* Participants are permitted to participate in another study or trial in addition to PRO-DIGI

Exclusion Criteria:

* Non conversationaI standard of English
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing major abdominal surgery for gastrointestinal, urological, or gynaecological indications OR patients being treated for intestinal obstruction regardelss of aetiology.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Completion of interviews (stage one) | Within one month of treatment
  completions of interview by group 1
Completion of questionnaire (stage three) | Within two weeks of treatment
  completion of questionnaire by group 3
Completion of face validity assessment (stage two) | Within one month of treatment
  Assessment of face validity using the QQ-10 (Questionnaire quality-10 item) questionnaire by group 2

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Lee, PhD, Principal Investigator — University of Sheffied and Sheffield Teaching Hospitals
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised transcriptions of phase one interviews will be made available on our institution open access data repository. Other data relates to refinement of the PROM and is not relevant outside of this study.